CLINICAL TRIAL: NCT04207684
Title: Generation of Biological Samples Positive to Testosterone for Anti-doping Control
Acronym: TST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/TST
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
Keywords: Testosterone; Anti-doping control; Athletic performance
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testosterone (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 5 days after administration (6 fractions: 0-12h, 12-24h, 24-48h, 48-72h, 72-96h, 96-120h post-administration).
  Interventions: Drug: Testosterone injection

INTERVENTIONS:
Drug: Testosterone injection — 250 mg of testosterone cypionate (equivalent to 174,8 mg of testosterone) administered via intramuscular injection in a single dose (2 mL)
  Other Names: Testex Prolongatum® 250 mg/2 mL

SUMMARY:
Background:

Testosterone is a steroid widely known to improve physical performance due to its protein-anabolic effect. Like other androgenic anabolic steroids (EAA), testosterone is included on the World Anti-Doping Agency (WADA) list of prohibited substances.

EAA are the most detected banned substances in anti-doping controls. Therefore, different analytical strategies are required to improve its detection.

Hypothesis:

The intramuscular administration of 250 mg of testosterone (cypionate) in healthy subjects allows generating detectable concentrations of the drug in urine. Positive urine samples will enable to identify analytical strategies for doping control.

Objectives:

Primary objective: To measure the concentrations of testosterone in urine for anti-doping control samples.

Secondary objective: To identify metabolites and precursors of testosterone in urine. To assess safety and tolerability of the drug used.

Methods:

Phase I, open, non-randomized clinical trial, with a treatment condition (testosterone) administered via intramuscular injection to 4 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between 18 and 50 years.
* Able to understand and accept the trial procedures and able to sign an informed consent.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed before the test within normal limits. Minor or occasional variations of these limits will be allowed if, in the opinion of the Principal Investigator and taking into account the state of science, they have no clinical significance, do not pose a risk to the subject and do not interfere in the product evaluation. These variations and their non-relevance will be specifically justified in writing.
* Body mass index (weight/height^2) between 19 and 25 kg/m2 and weight between 50 and 90 kg. BMI between 25 and 27 kg/m2 may be included according to Principal Investigator's criteria.

Exclusion Criteria:

* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance or similar nonapeptides, or to any of the excipients.
* Patient with history or current presence of breast cancer, liver cancer, or suspicion or confirmation of prostate carcinoma.
* History or current presence of prostate syndrome symptoms: frequent urination (both day and night), difficulty in starting urination, weak or discontinuous urinary stream, feeling of incomplete bladder emptying, or benign prostatic hyperplasia diagnosis.
* Levels of prostate specific antigen (PSA) > 4 ng/mL.
* Hematocrit value >50%.
* Patients with acute abdominal pain of unknown origin.
* Clinical background or evidence of gastrointestinal, hepatic, renal disorder or others that may involve an alteration of the absorption, distribution, metabolism or excretion of the drug, or that are suggestive of gastrointestinal irritation by drugs.
* Clinical background or evidence of psychiatric disorders, alcoholism, drug abuse or habitual consumption of psychoactive drugs.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Having suffered some organic disease or major surgery in the six months prior to the start of the study.
* Clinical background or evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by him/her, may pose a risk to the subjects or may interfere with the objectives of the study. Especially history of venous thrombosis or thromboembolic disorders, thrombophilic alteration, edema, hypercalcemia, polycythemia, nephrosis, liver disease with altered liver function tests and porphyria.
* Having taken medication regularly in the month prior to the study sessions. Treatment with single doses of symptomatic medication in the week prior to the study sessions will not be a reason for exclusion if it is assumed that the drug has been completely eliminated on the day of the experimental session.
* Smokers of more than 20 cigarettes a day in the 3 months before the study.
* Consumption of more than 40 g of alcohol daily.
* Consumers of more than 5 coffees, teas, cola drinks, or other stimulant drinks or with xanthines daily in the 3 months prior to the study start.
* Being unable to understand the nature, consequences of the trial and the procedures that are asked to follow.
* Positive serology for hepatitis B, C or HIV.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Urine concentration of testosterone | 0-12 hours post-administration (Day 1)
  Concentration of testosterone in fraction-1 urine samples
Urine concentration of testosterone | 12-24 hours post-administration (Day 1)
  Concentration of testosterone in fraction-2 urine samples
Urine concentration of testosterone | 24-48 hours post-administration (Day 2)
  Concentration of testosterone in fraction-3 urine samples
Urine concentration of testosterone | 48-72 hours post-administration (Day 3)
  Concentration of testosterone in fraction-4 urine samples
Urine concentration of testosterone | 72-96 hours post-administration (Day 4)
  Concentration of testosterone in fraction-5 urine samples
Urine concentration of testosterone | 96-120 hours post-administration (Day 5)
  Concentration of testosterone in fraction-6 urine samples

SECONDARY OUTCOMES:
Urine concentration of testosterone metabolites | 0-12 hours post-administration (Day 1)
  Concentration of testosterone metabolites in fraction-1 urine samples
Urine concentration of testosterone metabolites | 12-24 hours post-administration (Day 1)
  Concentration of testosterone metabolites in fraction-2 urine samples
Urine concentration of testosterone metabolites | 24-48 hours post-administration (Day 2)
  Concentration of testosterone metabolites in fraction-3 urine samples
Urine concentration of testosterone metabolites | 48-72 hours post-administration (Day 3)
  Concentration of testosterone metabolites in fraction-4 urine samples
Urine concentration of testosterone metabolites | 72-96 hours post-administration (Day 4)
  Concentration of testosterone metabolites in fraction-5 urine samples
Urine concentration of testosterone metabolites | 96-120 hours post-administration (Day 5)
  Concentration of testosterone metabolites in fraction-6 urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Aldea Perona, Dr, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No